CLINICAL TRIAL: NCT00003018
Title: A Phase II Trial of Infusional 5-Fluorouracil (5-FU), Calcium Leucovorin (LV), Mitomycin-C (Mito-C), and Dipyridamole (D) in Patients With Locally Advanced Unresected Pancreatic Adenocarcinoma
Brief Title: S9700 Combination Chemotherapy in Treating Patients With Stage II or Stage III Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000065599; S9700 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2004-04-22 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2013-01

CONDITIONS: Pancreatic Cancer
Keywords: stage II pancreatic cancer; stage III pancreatic cancer; duct cell adenocarcinoma of the pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Dipyridamole; Fluorouracil; Leucovorin; Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemotherapy (Experimental): dipyridamole: 75mg/dose, PO, Days 1-28 of 5 week cycle; fluorouracil: 200 mg/m^2/day, continuous IV, Days 1-28 of 5 week cycle; leucovorin calcium: 30 mg/m^2/day, IV, Days 1,8,15,22 of 5 week cycle; mitomycin C: 10 mg/m^2, IV, Day 1 of 6 week cycle (for only 4 cycles)
  Interventions: Drug: dipyridamole; Drug: fluorouracil; Drug: leucovorin calcium; Drug: mitomycin C

INTERVENTIONS:
Drug: dipyridamole — 75mg/dose, PO, Days 1-28 of 5 week cycle
  Other Names: Persantine; NSC-515776
Drug: fluorouracil — 200 mg/m^2/day, continuous IV, Days 1-28 of 5 week cycle
  Other Names: 5-fluorouracil; 5-FU; NSC-19893
Drug: leucovorin calcium — 30 mg/m^2/day, IV, Days 1,8,15,22 of 5 week cycle
  Other Names: NSC-3590
Drug: mitomycin C — 10 mg/m^2, IV, Day 1 of 6 week cycle (for only 4 cycles)
  Other Names: Mutamycin; NSC-26980

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. Chemotherapy following surgery may be an effective treatment for pancreatic cancer.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy in treating patients with stage II or stage III pancreatic cancer that has not been surgically removed.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the one year overall survival rate of patients with advanced, unresectable pancreatic cancer treated with fluorouracil, leucovorin, mitomycin and dipyridamole. II. Assess the response rate in this group of patients. III. Evaluate the frequency and severity of the toxic effects associated with this therapy. IV. Assess the rate of resectability in patients who respond to therapy.

OUTLINE: All patients undergo surgical placement of an indwelling central venous line. Patients receive fluorouracil IV by continuous infusion on days 1-28, leucovorin calcium IV on days 1, 8, 15, and 22, oral dipyridamole on days 1-28, and mitomycin IV every 6 weeks starting on day 1. Treatment repeats every 6 weeks for 4 courses. Patients with a partial or complete response are reevaluated for possible surgical resection. Resected patients resume chemotherapy 4-8 weeks after surgery for an additional 16 weeks. Patients are followed every 6 months for 2 years, then annually until death.

PROJECTED ACCRUAL: A total of 55 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically proven stage II or III pancreatic adenocarcinoma Ductal adenocarcinoma Mucinous noncystic carcinoma Signet ring cell carcinoma Adenosquamous carcinoma Undifferentiated (anaplastic) carcinoma Mixed ductal-endocrine carcinoma Well differentiated adenocarcinoma Moderately well or poorly differentiated adenocarcinoma Undifferentiated ductal carcinoma Must have unresectable and localized disease Measurable or evaluable disease

PATIENT CHARACTERISTICS: Age: Not specified Performance status: SWOG 0-2 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: Not pregnant or nursing Fertile patients must use effective contraception Loss of no greater than 15% of actual body weight Oral intake of greater than 1,200 calories per day No other malignancy within the past 5 years except adequately treated basal or squamous cell skin cancer, carcinoma in situ of the cervix, or any stage I or II cancer that is currently in complete remission

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior systemic chemotherapy for pancreatic cancer Endocrine therapy: Not specified Radiotherapy: No prior radiation therapy for pancreatic cancer Surgery: At least 2 weeks since prior surgical bypass procedure and recovered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 1997-09; Primary Completion 2002-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Overall Survival | One year

SECONDARY OUTCOMES:
Response rate in patients with measurable disease | From date of registration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
Toxicities | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
Resectability of patents who respond to this regimen | From date of registration until the date of patients achieving complete or partial response assessed up to 100 months

CONTACTS AND LOCATIONS:
Overall Officials: William H. Isacoff, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (84):
- United States (84):
  - MBCCOP - University of South Alabama, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Beckman Research Institute, City of Hope, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Medical Center, Sacramento, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - Oregon Cancer Center at Oregon Health Sciences University, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Texas Tech University Health Science Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington

REFERENCES:
- [Result] Isacoff WH, Bendetti JK, Barstis JJ, Jazieh AR, Macdonald JS, Philip PA. Phase II trial of infusional fluorouracil, leucovorin, mitomycin, and dipyridamole in locally advanced unresectable pancreatic adenocarcinoma: SWOG S9700. J Clin Oncol. 2007 May 1;25(13):1665-9. doi: 10.1200/JCO.2006.06.7637. PMID 17470859
- [Result] Isacoff WH, Benedetti J, MacDonald JS, et al.: Continuous infusion (CI) 5 fluorouracil (5FU), leucovorin (LV), mitomycin C (Mito C) and dipyridamole (D) in patients with locally advanced unresectable pancreatic adenocarcinoma - a phase II trial of the Southwest Oncology Group. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-544, 2002.